CLINICAL TRIAL: NCT00614705
Title: A Four Week, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 2A Study Of PH-797804 In The Treatment Of Post-Herpetic Neuralgia
Brief Title: PH-797804 Versus Placebo For The Treatment Of Neuropathic Pain Associated With Post-Herpetic Neuralgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trials Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A6631013
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Neuralgia, Postherpetic
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — PH 797804

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: PH-797804
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PH-797804 — 6 mg dose in oral capsule form, once daily for 28 days
  Arms: 1
Drug: Placebo — oral capsule form, once daily for 28 days
  Arms: 2

SUMMARY:
This is a proof-of-concept study to determine if PH-797804 reduces neuropathic pain associated with post-herpetic neuralgia. Suitable patients will be randomized to receive either PH-797804 or placebo for 4 weeks, during which time they will also record their pain symptoms using various pain scales.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age
* Patients must have pain present for more than 3 months after healing of the Herpes zoster skin rash. There is no upper limit on the duration of PHN.
* Patients at screening visit (V1) must have a score ≥40 mm on the Pain Visual Analog Score (VAS).

Exclusion Criteria:

* Patients having other severe pain, which may impair the self-assessment of the pain due to post-herpetic neuralgia
* History within the previous year of: myocardial infarction, cardiac arrhythmia (e.g. atrial fibrillation, paroxysmal atrial fibrillation, atrial flutter, supraventricular tachycardia, ventricular tachycardia), left ventricular failure, New York Heart Association (NYHA) Class III-IV congestive heart failure requiring treatment, unstable angina, coronary angioplasty, coronary artery bypass grafting (CABG) or cerebrovascular accident (including transient ischemic attacks).
* Tuberculosis without treatment and/or positive tuberculin reaction to PPD (Purified Protein Derivative) without known (documented) vaccination with the bacilli Calmette-Guerin vaccine (BCG).
* A positive approved immunoassay/ELISA blood test for TB (e.g. TB T-SPOT™, QuantiFERON-Gold
* Any clinically significant skin lesions as described in Common Terminology Criteria for Adverse Events for Dermatology (CTCAE) Version 3.0
* ECG abnormalities at screening or randomization
* Evidence of organ dysfunction or hematopoietic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-04; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline to endpoint in weekly average pain score using the 11-point daily pain rating scale | 4 weeks

SECONDARY OUTCOMES:
PH-797804 pharmacokinetics | Weeks 1, 2, and 4
Patient global impression of change | Week 4
Neuropathic Pain Symptom Inventory | Baseline and Weeks 1, 2, and 4

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (21):
- Pfizer Investigational Site, Viña del Mar, Región de Valparaíso, Chile
- Russia (3):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
  - Pfizer Investigational Site, Yaroslavl
- Spain (5):
  - Pfizer Investigational Site, Cadiz, Cadiz
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Ourense, Ourense
  - Pfizer Investigational Site, Seville, Sevilla
  - Pfizer Investigational Site, Valencia, Valencia
- Sweden (2):
  - Pfizer Investigational Site, Linköping
  - Pfizer Investigational Site, Stockholm
- Ukraine (6):
  - Pfizer Investigational Site, Dnipropetrovsk
  - Pfizer Investigational Site, Donetsk
  - Pfizer Investigational Site, Kharkiv
  - Pfizer Investigational Site, Kyiv
  - Pfizer Investigational Site, Odesa
  - Pfizer Investigational Site, Simferopol
- United Kingdom (4):
  - Pfizer Investigational Site, Bexhill-on-Sea, East Sussex
  - Pfizer Investigational Site, Blackpool, Lancashire
  - Pfizer Investigational Site, Weybridge, Surrey
  - Pfizer Investigational Site, Solihull

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6631013&StudyName=PH-797804%20Versus%20Placebo%20For%20The%20Treatment%20Of%20Neuropathic%20Pain%20Associated%20With%20Post-Herpetic%20Neuralgia